CLINICAL TRIAL: NCT05652036
Title: Procedural Discomfort Related to Number of Intradetrusor Injections of OnabotulinumtoxinA for Idiopathic Overactive Bladder: A Randomized Control Trial of an Alternate Reconstitution Volume and Injection Template Protocol
Brief Title: Procedural Discomfort Related to Number of Intradetrusor Botox Injections
Acronym: BIND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rose Khavari, M.D., Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00028592
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Urinary urgency; Urgency incontinence; Botox
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 5 mL Group (Active Comparator): 100 units BTX-A reconstituted in 5 mL normal saline, injected into the bladder in 5 separate injections of 1 mL. One injection will be at the trigone.
  Interventions: Biological: Intradetrusor Botox Injections
- 10 mL Group (Active Comparator): 100 units BTX-A reconstituted in 10 mL normal saline, injected into the bladder in 10 separate injections of 1 mL. One injection will be at the trigone
  Interventions: Biological: Intradetrusor Botox Injections

INTERVENTIONS:
Biological: Intradetrusor Botox Injections — 100 units of OnabotuliumtoxinA is injected into the detrusor muscle in 1 mL aliquots using a cystoscope.

SUMMARY:
Injection of intradetrusor OnabotulinumtoxinA (BTX-A) is a highly efficacious therapy with a reliable safety profile and demonstrable improvements in subjective and objective measures for overactive bladder (OAB) symptom control. This procedure can be performed in the office with an evidence-based standard dosing of 100 units for idiopathic OAB. This is a single-blinded, randomized control trial is to evaluate and optimize the technique for performing intradetrusor injections of BTX-A for idiopathic OAB. This trial proposes two different reconstitution and injection schema to study patient-centered outcomes related to procedural discomfort and symptom relief.

DETAILED DESCRIPTION:
This will be a single-blinded, parallel randomized control trial (RCT) utilizing two study arms. This trial will be designed and reported as outlined in the CONSORT guidelines

The primary aim of this study is to evaluate perceived discomfort using the Numeric Pain Scale (NPS) during office injection of intradetrusor BTX-A via two different injection techniques and reconstitution volumes.

The secondary aims of this study are to evaluate treatment effectiveness and patient satisfaction of treatment with BTX-A using validated questionnaires. Investigators will also compare procedure time and post-procedure complication rates between the two study groups.

Study Groups: The patients will be randomized in a 1:1 fashion to one of two groups:

* 100 units BTX-A reconstituted in 5 mL normal saline, injected into the bladder in 5 separate injections of 1 mL. One injection will be at the trigone
* 100 units BTX-A reconstituted in 10 mL normal saline, injected into the bladder in 10 separate injections of 1 mL. One injection will be at the trigone

The primary outcome will be measured on the day of the procedure using the NPS scale. Investigators will follow up with patients at 30 days post-procedure to assess treatment effectiveness, overall satisfaction, and post-procedure outcomes using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled to undergo 100 units intradetrusor BTX-A injections in the office for the diagnosis of idiopathic overactive bladder within the departments of Urology and Urogynecology
* 18 years of age or older
* Able to give informed consent in English or Spanish
* Understand and are willing to undergo follow-up and complete all questionnaires as described in this protocol

Exclusion Criteria:

* Neurogenic bladder related to prior diagnosis of neurological conditions such as cerebral vascular accident within 6 months prior to treatment, Parkinson's Disease, Multiple Sclerosis, myelomeningocele, traumatic neurologic or spinal injury, or idiopathic diagnosis of neurogenic bladder.
* Symptomatic UTI at the time of procedure, defined as positive nitrites or high-volume leukocyte esterase on urine dip in addition to at least one of the following symptoms: dysuria, gross hematuria, suprapubic pain, frequency/urgency above baseline
* Diagnosis of a bladder pain syndrome or other chronic pain syndromes including fibromyalgia, chronic pelvic pain, pelvic floor dysfunction, levator myalgia
* Known bladder malignancy
* Previous history of bladder augmentation or reconstructive surgery not related to prolapse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose Khavari, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miceli LM, Antosh DD, Nisar T, Stewart J, Rutledge EC, Khavari R. Pain Related to Intradetrusor BotulinumtoxinA: A Randomized Clinical Trial. Urogynecology (Phila). 2024 Mar 1;30(3):337-344. doi: 10.1097/SPV.0000000000001487. PMID 38484251

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 mL Group | 10 mL Group
Started | 52 | 56
Completed | 52 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mL Group | 10 mL Group | Total
Number analyzed (Participants) | 52 | 56 | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (14.3) | 70.6 (10.3) | 67.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 56 | 108
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 46 | 45 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Medical Co-Morbidities [Count of Participants; unit: Participants]
  Diabetes | 9 | 8 | 17
  Depression | 23 | 18 | 41
  Neurologic Diagnosis | 15 | 10 | 25
  Recurrent Urinary Tract Infection | 5 | 12 | 17
Surgical History [Count of Participants; unit: Participants]
  Hysterectomy | 23 | 35 | 58
  Prolapse Repair | 16 | 10 | 26
  Incontinence Procedure | 14 | 6 | 20
First Botox Injection [Count of Participants; unit: Participants]
  Yes | 22 | 20 | 42
  No | 30 | 36 | 66

OUTCOME MEASURES:

1. Primary Outcome: Participant Discomfort Related to BTX-A Injection
Description: Participants will assess their discomfort using the Numeric Pain Scale (NPS), a validated 11-point scale (0-10) where higher scores indicate greater pain, before and immediately after the procedure. Procedural discomfort will be evaluated by comparing the change in NPS scores from pre- to post-procedure between study groups.
Time Frame: Immediately post-procedure (up to 45min after intradetrusor BTX-A injections)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5 mL Group | 10 mL Group
Number analyzed (Participants) | 52 | 56
score on a scale | 3.2 (2.3) | 3.6 (2.1)
Statistical Analysis 1: Comparison: 5 mL Group vs 10 mL Group; Difference in NPS score pre- and post-procedure; Test type: Other; p = 0.21, t-test, 2 sided — Threshold for statistical significance used P-value <0.05

2. Secondary Outcome: Procedural Efficacy - Overactive Bladder Questionnaire Short-Form (OAB-q SF)
Description: Efficacy will be evaluated using the Overactive Bladder Questionnaire Short-Form (OAB-q SF), a validated instrument designed to measure symptom bother (SB) and the impact of OAB on health-related quality of life (HRQL). This questionnaire is administered on the day of the procedure (baseline) and again 30 days post-procedure. Changes in SB and HRQL scores assess improvement in OAB symptoms following BTX-A treatment.
  The OAB-q SF includes 19 items divided into two subscales: a 6-item SB scale (Questions 1-6) and a 13-item HRQL scale (Questions 7-19). SB items are scored from 1 ("not at all") to 6 ("a very great deal"), yielding a total SB score range of 6 to 36, with higher scores indicating greater symptom bother. HRQL items are scored from 1 ("none of the time") to 6 ("all of the time"), with total scores ranging from 13 to 78, where higher scores reflect better quality of life.
  We report here the mean change in SB and HRQL scores from baseline to 30 days post-treatment.
Time Frame: Prior to BTX-A injections and 30 days post-procedure
Population: Follow-up data 30-days post-treatment was obtained from 69% (n = 36) of participants in the 5 mL/5 injection arm and 77% (n = 43) of participants in the 10 mL/10 injection arm.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | 5 mL Group | 10 mL Group
Number analyzed (Participants) | 36 | 43
Units on a scale
  OAB-q SF (SB (mean difference)) | -22.4 [-93 to 73] | -38.1 [-100 to 60]
  OAB-q SF (HRQL (mean difference)) | 14.59 [-59 to 60] | 26.24 [-30 to 71]
Statistical Analysis 1: Comparison: 5 mL Group vs 10 mL Group; Difference in overactive bladder symptom bother before and after treatment; Test type: Other; p = .07, t-test, 2 sided — Threshold for statistical significance used P-value <0.05
Statistical Analysis 2: Comparison: 5 mL Group vs 10 mL Group; Difference in overactive bladder HRQL mean before and after treatment; Test type: Other; p = 0.16, t-test, 2 sided — Threshold for statistical significance used P-value <0.05

3. Secondary Outcome: Overall Treatment Satisfaction
Description: Overall treatment satisfaction will be assessed at 30-days post-procedure via a "yes or no" response to inquiry about overall satisfaction with the procedure and results of their BTX-A treatment
Time Frame: 30 days post-procedure
Population: Thirty-day follow-up data were available for 69% (n = 36) in the 5 mL/5 injection arm and 77% (n = 43) in the 10 mL/10 injection arm.
Measure: Count of Participants; unit: Participants
Groups:
- 5ml/ 5 Injection: Group of participants who received the least amount of injections
- 10ml/ 10 Injections: Group of participants who received the most injections
Arm/Group | 5ml/ 5 Injection | 10ml/ 10 Injections
Number analyzed (Participants) | 36 | 43
Participants
  Satisfied | 33 | 34
  Not Satisfied | 3 | 9
Statistical Analysis 1: Comparison: 5ml/ 5 Injection vs 10ml/ 10 Injections; Participant rated procedural satisfaction assessed 30-days post-procedure; Test type: Other; p = 0.21, Chi-squared

4. Secondary Outcome: Impression of Clinical Improvement
Description: Patients impression of clinical improvement after treatment will be assessed at 30-day post-procedure via the Clinical Global Impression - Improvement Scale (CGI-I). The CGI-I is a seven point verbal scale with higher values indicating higher impression of symptomatic improvement related to the treatment. Scale reports values as: Very much improved, Much improved, Minimally improved, No difference.
Time Frame: 30 days post-procedure
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mL Group | 10 mL Group
Number analyzed (Participants) | 36 | 43
Participants
  Very much improved | 9 | 9
  Much improved | 18 | 16
  Minimally improved | 7 | 15
  No difference | 2 | 3
Statistical Analysis 1: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Clinical Global Impression of Improvement scale sores reported by participants as very much improved after treatment; p = 0.79, Chi-squared
Statistical Analysis 2: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Clinical Global Impression of Improvement scale sores reported by participants as much improved after treatment; p = 0.27, Chi-squared
Statistical Analysis 3: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Clinical Global Impression of Improvement scale sores reported by participants as minimally improved after treatment; p = 0.14, Chi-squared
Statistical Analysis 4: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Clinical Global Impression of Improvement scale sores reported by participants as no difference after treatment; p = 1.0, Chi-squared

5. Secondary Outcome: Procedural Outcomes
Description: We will review the electronic medical record to evaluate instances of symptomatic urinary tract infection, bothersome incomplete bladder emptying requiring catheterization, and instances of bleeding requiring evaluation after the procedure.
Time Frame: 30 days post-procedure
Population: Post-procedural Adverse Outcomes - Urinary retention, Urinary tract infection, Bleeding requiring evaluation, Hematuria, Bladder pain, and Emergency department evaluation. n=36 and n=43 participants were evaluated for the 5ml and 10ml arms respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mL Group | 10 mL Group
Number analyzed (Participants) | 36 | 43
Participants
  Urinary retention | 0 | 2
  Urinary tract infection | 5 | 2
  Bleeding requiring evaluation | 0 | 0
  Hematuria | 1 | 0
  Bladder pain | 0 | 1
  Emergency department evaluation | 0 | 2
Statistical Analysis 1: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Rates of urinary retention observed in participants after BTX-A treatment; p = 0.5, Chi-squared
Statistical Analysis 2: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Rates of urinary tract infection observed in participants after BTX-A treatment; p = 0.24, Chi-squared
Statistical Analysis 3: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Rates of bleeding requiring evaluation observed in participants after BTX-A treatment; p = 1.0, Chi-squared
Statistical Analysis 4: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Rates of hematuria observed in participants after BTX-A treatment; p = 0.46, Chi-squared
Statistical Analysis 5: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Rates of bladder pain observed in participants after BTX-A treatment; p = 1.0, Chi-squared
Statistical Analysis 6: Comparison: 5 mL Group vs 10 mL Group; Test type: Other — Rates of ER department evaluations observed in participants after BTX-A treatment; p = 0.5, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 month post-treatment
Description: Thirty-day AE data were available for 69% (n = 36) of participants in the 5 mL/5 injection arm and 77% (n = 43) of participants in the 10 mL/10 injection arm.
Arm/Group | 5 mL Group | 10 mL Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/43
Other Adverse Events (participants affected / at risk) | 6/36 | 7/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mL Group (N=36) | 10 mL Group (N=43)
Urinary Tract Infection (Renal and urinary disorders) | 5 (5) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Bleeding Requiring Evaluation (Renal and urinary disorders) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Emergency Department Evaluation (Renal and urinary disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Possible small variations in injection technique were minimized through physician training. Patients were blinded to treatment, but non-naive patients may have biased pain scores based on prior experiences. Loss to follow-up at 30 days limits conclusions on secondary outcomes related to patient experience and procedural efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT05652036/Prot_SAP_001.pdf